CLINICAL TRIAL: NCT05252403
Title: Measurable Residual Disease Driven Strategy for One or Two Infusions of Non- Viral, Transposon-manipulated CARCIK (CD19) Cells: A Phase II Study in Pediatric and Adult Patients With Relapsed/Refractory B Cell Precursor ALL (BCP-ALL)
Brief Title: Residual Disease Driven Strategy for CARCIK (CD19) in Adults/Pediatric BCP-ALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Matilde Tettamanti Menotti De Marchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT03CARCIK
Record Dates: First submitted 2022-01-24; First posted 2022-02-23 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARCIK-CD19 (Experimental)
  Interventions: Genetic: PTG-CARCIK-CD19

INTERVENTIONS:
Genetic: PTG-CARCIK-CD19 — PTG-CARCIK-CD19 cells is a gene therapy medicinal product (GTMP) composed of genetically modified allogeneic T lymphocytes formulated as cell suspension in normal saline solution and freezing media

SUMMARY:
This is a single arm, open-label, multi-center, phase II study to determine the activity and the safety of a therapeutic strategy that allows a second CARCIK-CD19 cells infusion, driven by the status of disease from one month after the first infusion, in adult and pediatric patients with r/r BCP- ALL.

ELIGIBILITY:
Inclusion Criteria:

Children (1-17) and adults (18-75 years old);

* Relapsed or refractory adult and pediatric B- ALL as defined for the presence of bone marrow with ≥ 5% lymphoblasts by morphologic assessment, or if <5%, with at least 1% of molecular disease at PCR;
* Evidence of CD19 tumor expression in bone marrow and/or peripheral blood by flow cytometry;
* Diagnosis of CD19 positive ALL in the bone marrow, and/or peripheral blood and/or extramedullary sites with the exclusion of Central Nervous System (CNS) if CNS-3 disease.

Exclusion Criteria:

* GVHD Grades II-IV for patients who had previously been transplanted; 2. Any cell therapy in the previous 30 days;
* Patient with concomitant life-threatening infectious disease;
* Lansky/Karnofsky score <60;
* Patients with hepatic or renal disease as specific above;
* Pregnant or breast-feeding females;
* Rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy;

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the overall response rate: change from baseline at day 28 after the first CARCIK-CD19 infusion | Baseline and day 28
  At baseline and at Day 28 after infusion: lymphoblasts < 5% at morphological evaluation of bone marrow aspirate
To evaluate the overall response rate: change from baseline at day 28 after the first CARCIK-CD19 infusion | Baseline and day 28
  At baseline and at Day 28 after infusion: lymphoblasts < 5% at flow cytometry bone marrow evaluation
To evaluate the overall response rate: change from baseline at day 28 after the first CARCIK-CD19 infusion | Baseline and day 28
  At baseline and at Day 28 after infusion: molecular evaluation of disease positivity <0.01%
To evaluate the duration of response of patients treated with CARCIK - CD19 cells. Change from day 28 at month 2, 3, 4, 5, 6, 9 and 12 | Day 28 and month 2, 3, 4, 5, 6, 9 and 12
  Day 28 and month 2, 3, 4, 5, 6, 9 and 12: lymphoblasts < 5% at morphological evaluation of bone marrow aspirate
To evaluate the duration of response of patients treated with CARCIK - CD19 cells. Change from day 28 at month 2, 3, 4, 5, 6, 9 and 12 | Day 28 and month 2, 3, 4, 5, 6, 9 and 12
  Day 28 and month 2, 3, 4, 5, 6, 9 and 12: lymphoblasts < 5% at flow cytometry bone marrow evaluation
To evaluate the duration of response of patients treated with CARCIK - CD19 cells. Change from day 28 at month 2, 3, 4, 5, 6, 9 and 12 | Day 28 and month 2, 3, 4, 5, 6, 9 and 12
  Day 28 and month 2, 3, 4, 5, 6, 9 and 12: molecular evaluation of disease positivity <0.01%

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale PG23, Bergamo
  - Fondazione MBBM, Monza

IPD SHARING:
Plan to Share IPD: No